CLINICAL TRIAL: NCT00684957
Title: Differential Effects of rhGH vs. rhIGF-1 on Cardiovascular Risk Factors in Adult Patients With Growth Hormone Deficiency
Brief Title: Differential Effects of rhGH vs. rhIGF-1 on Cardiovascular Risk Factors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: Tercica (Industry)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine at the Columbia University Medical Center, Dept of Medicine Endocrinology, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAC2883; Tercica-001 (Other: Tercica)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Growth Hormone Deficiency
Keywords: rhGH; rhIGF-1
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recombinant Human Growth Hormone first (Active Comparator): Subjects will take rhGH for eight weeks followed by a two month wash out period and then will cross over to rhIGF1 for eight weeks.
  Interventions: Drug: Recombinant Human Growth Hormone; Drug: Recombinant Human IGF-1
- Recombinant Human IGF-1 (Active Comparator): Subjects will take rhIGF1 for eight weeks followed by a two month wash out period and then will cross over to rhGH for eight weeks.
  Interventions: Drug: Recombinant Human Growth Hormone; Drug: Recombinant Human IGF-1

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone — 300 mcg sc qd (which may be increased to 400 mcg sc qd after 4 weeks)
  Other Names: rhGH
Drug: Recombinant Human IGF-1 — 30 µg/kg for first 4 weeks (may be increased thereafter based on IGF-1 levels)
  Other Names: rhIGF-1

SUMMARY:
The purpose of this study is to see if giving growth hormone or insulin-like growth factor-1 (IGF-1) to subjects with growth hormone deficiency effects cardiovascular risk factors differently.

DETAILED DESCRIPTION:
Insulin-like growth factor-1 (IGF-1) in some circumstances acts as the mediator of the metabolic effects of growth hormone. However, there is some evidence to suggest that growth hormone (GH) and IGF-1 act differently in some metabolic pathways. We will study the differences between GH and IGF-1 when provided as therapy for growth hormone deficiency in adults. Specifically we will be assessing if either medication impacts cardiovascular risk factors and if so do they impact risk factors differently. Ten adult males ages 18-65 who are growth hormone deficient on stable medications and with stable magnetic resonance imaging (MRI) findings (in the event of a known pituitary mass) will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult male age 25-65 with documented growth hormone deficiency on stable doses x 3 months (at least) of any hormone replacement therapies and with stable MRIs x 2 years in the setting of a known pituitary mass.

Exclusion Criteria:

* Female gender
* current GH use or GH use within three months of the study
* diabetes
* hypoglycemia
* liver or kidney disease
* use of drugs that could increase GH secretion (i.e. L-dopa)
* alcohol or substance abuse
* use of investigational drugs within four weeks of our study and use of supraphysiologic doses of steroids within the previous six months.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U. Freda, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, College of Physicians and Surgeons, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Growth Hormone First, Then Recombinant Human IGF-1: Subjects will take Recombinant Human Growth Hormone (rhGH) for eight weeks followed by a two month wash out period and then will cross over to Recombinant Human IGF-1 (rhIGF1) for eight weeks.
  rhGH dose: 300 mcg sc qd (which may be increased to 400 mcg sc qd after 4 weeks)
  rhIGF1 dose: 30 µg/kg for first 4 weeks (may be increased thereafter based on IGF-1 levels)
- Recombinant Human IGF-1 First, Then Recombinant Human Growth Hormone: Subjects will take Recombinant Human IGF-1 (rhIGF1) for eight weeks followed by a two month wash out period and then will cross over to Recombinant Human Growth Hormone (rhGH) for eight weeks.
  rhGH dose: 300 mcg sc qd (which may be increased to 400 mcg sc qd after 4 weeks)
  rhIGF1 dose: 30 µg/kg for first 4 weeks (may be increased thereafter based on IGF-1 levels)
Period: Overall Study
Arm/Group | Recombinant Human Growth Hormone First, Then Recombinant Human IGF-1 | Recombinant Human IGF-1 First, Then Recombinant Human Growth Hormone
Started | 2 | 3
Completed | 0 | 2
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Subjects: Includes all subjects enrolled into the study.
Arm/Group | Study Subjects
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Serum Risk Markers Including Lipids, IL-6, CRP and Homocysteine
Time Frame: 2 months
Population: Levels of cardiovascular serum risk markers were not measured and thus not analyzed due to poor enrollment.
Arm/Group | Study Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in Visceral Adiposity, Intrahepatic and Intramyocellular Lipids
Time Frame: 2 months
Population: Visceral adiposity, intrahepatic and intramyocllular lipids were not measured/collected and thus not analyzed due to poor enrollment.
Arm/Group | Study Subjects
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Endothelial Cell Function
Time Frame: 2 months
Population: Endothelial cell function was not measured/collected and thus not analyzed due to poor enrollment.
Arm/Group | Study Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Recombinant Human Growth Hormone First, Then Recombinant Human IGF-1 | Recombinant Human IGF-1 First, Then Recombinant Human Growth Hormone
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes